CLINICAL TRIAL: NCT06234813
Title: Targeting TFPI With Concizumab to Improve Haemostasis in Glanzmann Thrombasthenia Patients: an in Vitro Study
Acronym: GLAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2021/44
Record Dates: First submitted 2023-03-21; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-09

CONDITIONS: Glanzmann Thrombasthenia
Keywords: Concizumab; Hemostatic capacity; Glanzmann Thrombasthenia
MeSH Terms: conditions — Thrombasthenia | interventions — Thromboplastin; Collagen; concizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glanzmann Thrombasthenia Group (Experimental): Patient with a clear diagnosis of Glanzmann Thrombasthenia, whatever the subtype of disease
  Interventions: Other: Clot formation in whole blood under flow in a microfluidic flow chamber coated with tissue factor and collagen; Other: : PRP viscoelastic changes under clot formation measured by thromboelastometry using RoTEM; Other: Thrombin Generation Assay (TGA) in PRP using TF trigger; Other: Global fibrinolytic capacity in PRP using reagents for in vitro triggering of the clot and its lysis; Other: Concizumab
- Healthy donors (Active Comparator): Healthy donor without haemorrhagic ant thrombotic medical history
  Interventions: Other: Clot formation in whole blood under flow in a microfluidic flow chamber coated with tissue factor and collagen; Other: : PRP viscoelastic changes under clot formation measured by thromboelastometry using RoTEM; Other: Thrombin Generation Assay (TGA) in PRP using TF trigger; Other: Global fibrinolytic capacity in PRP using reagents for in vitro triggering of the clot and its lysis

INTERVENTIONS:
Other: Clot formation in whole blood under flow in a microfluidic flow chamber coated with tissue factor and collagen — TTAS (single measurements)
  Clot formation in whole blood under flow (2000 s-1) in a microfluidic flow chamber coated with tissue factor and collagen (T-TAS with AR chip)
  1. 500 µL of whole blood for each point;
  2. 7 points for each condition;
  3. Around 4 mL of whole blood will be needed for each patient or healthy subject;
  4. Values for Area Under the Curve (Aritrary Unit), Occlusion Starting Time (min), Occlusion Time (min.) will be reported.
Other: : PRP viscoelastic changes under clot formation measured by thromboelastometry using RoTEM — ROTEM (single measurements)
  1. ROTEM cups will be added
     * 20 µL calcium reagent (STARTEM)
     * 20 µL of 2,940-fold prediluted r-ExTEM reagent (50,000 fold dilution relative to 340 µL in the cup) added
     * 300 µL spiked PRP at 250 G/L (2.5 mL of PRP/patient)
  2. Values for clot time (CT sec, clot formation time (CFT) sec, maximum clot formation (mm) will be reported.
Other: Thrombin Generation Assay (TGA) in PRP using TF trigger — TGA (single measurements)
  1. The following will be added to well:
     * 20 uL of PRP-Reagent
     * 80 uL of spiked PRP (600 µL/patient at 100 G/L)
     * 20 uL FluCa
  2. Values for thrombin activity versus time and the derived parameters incl. lag-time (min), time to peak (min), time to peak (min), ETP (Arbitrary Unit) will be reported.
Other: Global fibrinolytic capacity in PRP using reagents for in vitro triggering of the clot and its lysis — Global fibrinolytic capacity (Lysis Timer) in 100 µL of PRP (250 G/L) using reagents for in vitro triggering of the clot (thrombin and calcium) and its lysis (tissue-plasminogenactivator (t-PA). Around 1 mL of PRP in total Lysis time in min
Other: Concizumab — Thrombin generation assay (TGA), microchip flow-chamber assay (T-TAS, rotational thromboelastometry and global fibrinolytic capacity to investigate and compare the effects of mixing concizumab (200, 1000 and 4000 ng/mL) with the main bleed treatment options for persons with GT
  Arms: Glanzmann Thrombasthenia Group

SUMMARY:
Glanzmann thrombasthenia is a rare genetic disorder caused by the absence or the dysfunction of the main receptor present on the surface of platelets, integrin αIIbβ3 or GPIIb-IIIa.

The lack of this protein on the surface of platelets no longer allows these blood cells to bind to each other. This binding corresponds to the process of platelet aggregation.

Generally, local measures will control nasal and superficial bleeding whereas platelet transfusions are used to control or prevent life-threatening.

The main complication of this treatment is the risk of developing anti-αIIbβ3 antibodies directed against the absent protein and platelet transfusion therapy can become ineffective.

Activated recombinant factor VII (rFVIIa) provides an alternative treatment for GT patients who develop such antibodies. However, this therapy has a short duration of efficacy, requiring repeated intravenous administrations every 2 to 3 hours.

There is a new treatment, Concizumab, which has not yet been marketed. This treatment acts on TFPI (tissue factor pathway inhibitor). TFPI is a protein that occurs naturally in the body and prevents blood cells from binding to each other.

Concizumab works by blocking TFPI, which may allow sufficient clotting to prevent bleeding.

This treatment could replace recombinant activated factor VII (rFVIIa) because it has the advantage of a much longer duration of efficacy (about 3 days) and is administered subcutaneously.

DETAILED DESCRIPTION:
This is in vitro research. The treatment will be tested on blood samples. This will allow us to evaluate in vitro the ability of Concizumab to restore coagulation compared to the usual treatments of platelet transfusions and recombinant activated factor VII (rFVIIa).

This is a single-center study conducted at the Bordeaux University Hospital, which included 10 with Glanzmann thrombasthenia patients and 10 healthy donors over a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

Glanzmann Thrombasthenia Group:

* Patient ≥18 years old
* Patient with a clear diagnosis of Glanzmann Thrombasthenia (GT), whatever the subtype of disease
* Affiliated person or beneficiary of a social security scheme.
* Free, informed and written consent signed by the participant, and the investigator (at the latest on the day of inclusion and before any examination required by the research)

Control Group:

* Healthy donor ≥ 18 years old
* Healthy donor, without haemorrhagic ant thrombotic medical history
* Person should not work in the investigator's department.
* Affiliated person or beneficiary of a social security scheme
* Free, informed and written consent signed by the participant, and the investigator (at the latest on the day of inclusion and before any examination required by the research)

Exclusion Criteria:

For both patient groups:

* Patient who has taken aspirin or a nonsteroidal anti-inflammatory medication within the previous 10 days
* Patient who has received a platelet transfusion or recombinant activated factor VII hemostatic treatment within the previous 7 days
* Patient who participated in another interventional study involving a drug within 30 days of entering this protocol
* Psychiatric, social or behavioral condition judged to be non-compatible with the respect of the protocol
* Adult protected by the law

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Effects of mixing concizumab compared with the main bleed treatment options for persons with GT | One point at the inclusion
  The samples will be analysed by measurement of in vitro hemostatic capacity :
  * Clot formation in whole blood under flow (2000 s-1) in a microfluidic flow chamber coated with tissue factor and collagen. Values for Area Under the Curve (Aritrary Unit), Occlusion Starting Time (min), Occlusion Time (min.) will be reported
  * PRP viscoelastic changes under clot formation measured by thromboelastometry. Values for clot time (sec), clot formation time (sec), maximum clot formation (mm) will be reported
  * Thrombin Generation Assay in PRP using tissue factor trigger. Values for thrombin activity versus time and the derived parameters incl. lag-time (min.), time to peak (min), time to peak (min), ETP (Arbitrary Unit) will be reported
  * Global fibrinolytic capacity (Lysis Timer in min) in whole blood using reagents for in vitro triggering of the clot and its lysis

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu FIORE, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU Bordeaux - Laboratoire Hématologie, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No